CLINICAL TRIAL: NCT06138262
Title: Effectiveness of Preconception Nutrition Education for Prospective Brides to Prevent Anemia and Chronic Energy Deficiency During Pregnancy.
Brief Title: Preconception Nutrition Education Intervention for Prospective Brides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ratna Wulandari, Principal Investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2106769774
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: In this study there were 2 groups, namely the group that was given intervention and the group that was not given intervention / control group. The intervention group will be provided with education through a preconception nutrition education module and the leaflet, and the control group was given education using the leaflet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- health promotion education about preconception nutrition (Experimental)
  Interventions: Other: Health promotion of education pre-conception nutritional preparation

INTERVENTIONS:
Other: Health promotion of education pre-conception nutritional preparation — Providing education on pregnancy nutritional preparation during the preconception period 3 months before the wedding

SUMMARY:
This research focuses on the importance of preconception health care. In this research, an intervention was carried out providing health education regarding preconception nutritional preparation. Research methods used is a Quasi Experiment with the Non Equivalent Control Group method. Example used in this research were 100 prospective brides and grooms in Indonesia. The intervention group will be provided with education through a preconception nutrition education module and the brides health card, and the control group was given education using the brides health leaflet.

ELIGIBILITY:
Inclusion Criteria :

* Women aged 20 to 35 years old
* Have no history of disease that weakens anemia and nutritional intake
* Examination maximum 3 months before the wedding
* Prospective bridal couples do not delay the pregnancy program

Exclusion Criteria :

* Not complete premarital reproductive health examination

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Haemoglobin Level | one day
  Measurement of hemoglobin levels by taking a blood sample is then analyzed by laboratory staff at the health center (health facility service where the examination is carried out) then the results are written on the laboratory check results in units of measurement gr/dL with a normal value of at least 12 gr/dL with the subject being an adult woman and pregnant women in the 1st trimester..
Body Mass Index | one day
  Body mass index is measured by measuring body weight (kilograms) divided by height (meters) squared with units of measurement kg/m2 with subjects measured by adult women and pregnant women in the 1st trimester, with a minimum normal BMI value of 18.5 kg/m2.
Midupper Arm Circumference (MUAC) | one day
  MUAC is measured in adults women using a flexible meter line tape laid at the midpoint between the acromion and olecranon processes on the shoulder blade and the ulna, respectively, of the arm, with a normal value of at least 23.5 cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Puskesmas / Government First Level Health Facilities, Depok, West Java, Indonesia